CLINICAL TRIAL: NCT05577065
Title: A Randomised, Double-blinded, Placebo-controlled, Parallel Study, to Assess the Effect of a Probiotic on the Incidence, Duration and Severity of Upper Respiratory Tract Infections in Healthy Children
Brief Title: A Study to Assess the Effect of a Probiotic on Upper Respiratory Tract Infections in Healthy Children
Acronym: KLEENEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Archer-Daniels-Midland Company (Industry)
Collaborators: Atlantia Food Clinical Trials (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CTB2022TN108; AFCRO158 (Other: Atlantia Food Clinical Trials)
Record Dates: First submitted 2022-09-29; First posted 2022-10-13 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2024-11

CONDITIONS: Upper Respiratory Tract Infections; Upper Resp Tract Infection
Keywords: probiotic; microbiome
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: study consists of 2 arms, intervention and placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Experimental): Arm receiving investigational product (probiotic)
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Arm receiving placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Single strain probiotic in the form of a sachet with a daily dose of 3E+9 Colony Forming Unit (CFU) per day for 26 weeks.
  Arms: Active
Dietary Supplement: Placebo — Matching placebo in the form of a sachet once daily for 26 weeks
  Arms: Placebo

SUMMARY:
This study evaluates the efficacy of a single strain probiotic on the incidence, duration and severity of upper respiratory tract infections in healthy, school-age children.

ELIGIBILITY:
Inclusion Criteria:

1. Have a parent/guardian able to give written informed consent.
2. If ≥7 years, be able to give written informed assent.
3. Healthy children aged 2 - 8 years old.
4. In general good health, as determined by the investigator.
5. Attending a registered childcare provider or school.
6. Willing to consume the study product daily for the duration of the study.

Exclusion Criteria:

1. Has URTI symptoms at the time of randomisation.
2. Are <2 or ≥9 years old.
3. Diagnosed with concomitant chronic infections, chronic systemic diseases, autoimmune diseases (e.g. asthma - generally only formally diagnosed after child is 6 years), immunodeficiency, metabolic diseases, chronic respiratory tract diseases including respiratory allergies and cystic fibrosis or congenital cardiac defects.
4. Has a family household member that smokes cigarettes in the home.
5. Has taken antibiotics within the previous 2 weeks prior to randomisation.
6. Has taken probiotic supplements within the previous 2 weeks prior to randomisation
7. Daily intake of immune stimulating products, including but not limited to echinacea, vitamin C and zinc in the 2 weeks before randomisation (multivitamins allowed).
8. Has any significant health conditions that would prevent them from fulfilling the study requirements, put the Participant at risk or would confound the interpretation of the study results as judged by the investigator on the basis of medical history and routine laboratory test results.
9. Taking a medication that the investigator believes would interfere with the objectives of the study or pose a safety risk or confound the interpretation of the study results.
10. Has an active gastrointestinal disorder or previous gastrointestinal surgery (appendicectomy allowed).
11. Has a gastrointestinal or chronic infective disease (i.e., coeliac disease, diarrhoea, Crohn's disease, ulcerative colitis, irritable bowel syndrome, diverticulosis, stomach or duodenal ulcers, hepatitis, HIV, cancer, etc.), or with a history of such diseases.
12. Planned extensive travel (for >1 month) during the study duration.
13. Parent/guardian who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the study.
14. Participants may not be receiving treatment involving experimental drugs. If the Participant has been in a recent experimental trial/study, these must have been completed not less than 60 days prior to this study.
15. Any Participant who is the child of an employee of the study site or an Atlantia Clinical Trials employee or their close family member or a member of their household.

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-03-13 (Actual)

PRIMARY OUTCOMES:
Effect of 26 week consumption of probiotic on the total number of days that, otherwise healthy, children suffer from upper respiratory tract infection (URTI) | Entire follow up period (total of 180 days)
  Presence of an URTI defined by a score of >2 on the Jackson Cold Scale (maximum score 3) where a lower score means better outcomes compared to baseline

SECONDARY OUTCOMES:
Effect of 26 week consumption of probiotic on the number of children reporting at least one URTI | Day 0, Day 90, Day 180
  The presence of an URTI defined by a score of >2 on the Jackson Cold Scale (maximum score 3) where a lower score means better outcomes compared to baseline
Effect of 26 week consumption of probiotic on the average duration of URTIs reported by participants | Day 0, Day 90, Day 180
  Duration of URTI measured through the WURSS-K questionnaire (Maximum score 42) where a lower score means better outcomes compared to baseline
Effect of 26 week consumption of probiotic on the severity of URTI-related symptoms reported by participants | Day 0, Day 90, Day 180
  Severity of URTI measured through the WURSS-K questionnaire (Maximum score 42) where a lower score means better outcomes compared to baseline
Effect of 26 week consumption of probiotic on the total number of reported missed days of school/childcare due to illness | Day 0, Day 90, Day 180
  Recorded through the WURSS-K questionnaire (Maximum score 42) where a lower score means better outcomes compared to baseline
Effect of 26 week consumption of probiotic on the reported incidence of antibiotic use | Day 0, Day 90, Day 180
  Recorded through the WURSS-K questionnaire (Maximum score 42) where a lower score means better outcomes compared to baseline
Effect of 26 week consumption of probiotic on Salivary Immunoglobulin A levels (IgA) (mg/dL) | Day 0, Day 180
  Measured via saliva sample
Effect of 26 week consumption of probiotic on the incidence of gastrointestinal infections | Day 0, Day 90, Day 180
  Recorded through the WURSS-K questionnaire (Maximum score 42) where a lower score means better outcomes compared to baseline

OTHER OUTCOMES:
Faecal Microbiome analysis | Day 0, Day 180
  Shallow shotgun metagenomic sequencing for 20% of cohort

CONTACTS AND LOCATIONS:
Locations (1):
- Atlantia Food Clinical Trials, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No